CLINICAL TRIAL: NCT02355535
Title: (STM-03) Phase I Study of Procaspase Activating Compound-1 (PAC-1) in the Treatment of Advanced Malignancies - Component 1
Brief Title: Procaspase Activating Compound-1 (PAC-1) in the Treatment of Advanced Malignancies - Component 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanquish Oncology, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Oana Danciu, MD, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0057
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumor; Pancreatic Neuroendocrine Tumor; Neuroendocrine Tumors
Keywords: refractory; intolerant; solid tumors; PNET; neuroendocrine
MeSH Terms: conditions — Adenoma, Islet Cell; Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): Using a dose-escalation design, PAC-1 is administered orally on days 1-21, at the assigned dose, of a 28-day cycle.
  Interventions: Drug: PAC-1

INTERVENTIONS:
Drug: PAC-1 — PAC-1 is taken orally on days 1-21 of a 28-day cycle.
  Other Names: Procaspase Activating Compound-1

SUMMARY:
This Phase I dose escalation study will evaluate Procaspase Activating Compound-1 (PAC-1), a small molecule that activates procaspase -3 to caspase-3, resulting in apoptosis of cancer cells, in patients with advanced malignancies. As of March 1, 2019, only patients with neuroendocrine tumors will be enrolled in Component 1 of this study. PAC-1 is taken orally on days 1-21 of a 28-day cycle. The maximum tolerated dose (MTD) of PAC-1 (5 dose levels) will be determined using a modified-Fibonacci dose-escalation 3+3 design. Treatment continues until disease progression, unacceptable toxicity, physician discretion, or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Diagnosis of advanced solid tumor or hematologic malignancy (limited to lymphoma) that has failed or become intolerant to standard therapy
3. Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1, or lymphoma that fulfills the Deauville PET Criteria
4. Has an ECOG PS of 0, 1, or 2
5. Has total bilirubin < 1.5 mg/dL, serum albumin > 3.0 gm/dL, AST and ALT < 1.5 ULN or < 3 x ULN for subjects with known hepatic metastases
6. Has serum creatinine < 1.5 × ULN
7. Has hemoglobin ≥ 10 g/dL, ANC ≥ 1.5 × 109/L, and platelet count ≥ 100 × 109/L
8. Must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after capsule(s) administration
9. Must be willing and able to comply with study
10. Has read, understood, and signed the ICF
11. Women of childbearing potential must not be pregnant or breast-feeding. In addition, a medically acceptable method of birth control must be used or total abstinence. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP
12. Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male patients with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms at least one month after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative
13. Prior systemic treatments for metastatic disease are permitted but may not be ongoing, including targeted therapies, biologic response modifiers, chemotherapy, hormonal therapy, or investigational therapy
14. Willingness to donate blood for biomarker studies related to the type of therapies used in this trial and the tumor types being treated

Exclusion Criteria:

1. Had surgery within 4 weeks prior to study treatment except for minor procedures (hepatic biliary stent placement is allowed)
2. Gliomas are excluded, as well as any history of brain metastases, seizures or underlying brain injury
3. May not have received cytotoxic chemotherapy, targeted therapies, biologic response modifiers, chemotherapy, and hormonal therapy within the last 3 weeks, or nitrosureas within the last 6 weeks prior to study treatment.
4. Has a history of blood clots, pulmonary embolism, or DVT unless controlled by anticoagulant treatment
5. Has a history of an arterial thromboembolic event within the prior six months including CVA, TIA, MI, or unstable angina
6. Has uncontrolled HIV or hepatitis B or C
7. Has any clinically significant infection
8. Has any other severe, uncontrolled medical condition, including uncontrolled DM or unstable CHF
9. Radiation therapy to more than 25% of the bone marrow
10. Prior allogeneic bone marrow or organ transplantation
11. > Grade 1 peripheral neuropathy within 14 days before enrollment.
12. Patient has received other investigational drugs with 14 days before enrollment
13. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation
14. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinically significant (such as acute ischemia, left bundle branch block, ventricular arrhythmias) or baseline prolongation of the rate-corrected QT interval (e.g., repeated demonstration of QTc interval > 480 milliseconds)
15. Presence of any non-healing wound, fracture, or ulcer
16. Has any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance
17. Has any mental or medical condition that prevents the patient from giving informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 30 days post last dose
  The primary objective of this study component is to determine the maximum tolerated dose (MTD) of PAC-1 in patients with advanced, previously treated malignancy, by evaluation of toxicity and tolerability.

SECONDARY OUTCOMES:
Adverse Effects | Up to 30 days post final dose
  Characterize adverse effects (AE) of PAC-1 in patients with advanced malignancy.
Disease Response based on RECIST Criteria for patients with solid tumors | Up to 8 weeks following final dose
  Evaluate clinical response of PAC-1 in patients with solid tumors (RECIST v 1.1).
Disease Response based on Deauville PET Criteria for patients with lymphoma | Up to 8 weeks following final dose
  Evaluate clinical response of PAC-1 in patients with lymphoma (Deauville PET Criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Oana C Danciu, M.D., Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Regions Hospital, Saint Paul, Minnesota

REFERENCES:
- [Derived] Danciu OC, Holdhoff M, Peterson RA, Fischer JH, Liu LC, Wang H, Venepalli NK, Chowdhery R, Nicholas MK, Russell MJ, Fan TM, Hergenrother PJ, Tarasow TM, Dudek AZ. Phase I study of procaspase-activating compound-1 (PAC-1) in the treatment of advanced malignancies. Br J Cancer. 2023 Mar;128(5):783-792. doi: 10.1038/s41416-022-02089-7. Epub 2022 Dec 5. PMID 36470974